CLINICAL TRIAL: NCT02258555
Title: A Phase 1b Dose-escalation Study Evaluating the Safety, Pharmacodynamics, Pharmacokinetics, and Efficacy of GS-9901 in Subjects With Relapsed or Refractory Follicular Lymphoma, Marginal Zone Lymphoma, Chronic Lymphocytic Leukemia, or Small Lymphocytic Lymphoma
Brief Title: Safety, Pharmacodynamics, Pharmacokinetics, and Efficacy of GS-9901 in Adults With Relapsed or Refractory Follicular Lymphoma, Marginal Zone Lymphoma, Chronic Lymphocytic Leukemia, or Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-325-1348; 2014-005441-53 (EudraCT Number)
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Follicular Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Marginal Zone Lymphoma
Keywords: Chronic lymphocytic leukemia (CLL); Follicular lymphoma (FL); Small Lymphocytic Lymphoma (SLL); Phosphatidylinositol 3 kinase (PI3K); Marginal Zone Lymphoma (MZL)
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GS-9901 (Experimental): Participants will receive one of 6 escalating doses of GS-9901 once daily until unacceptable toxicity, substantial noncompliance, disease progression, pregnancy, initiation of another anti-cancer or experimental therapy, or other protocol-specified reasons for GS-9901 discontinuation.
  Interventions: Drug: GS-9901

INTERVENTIONS:
Drug: GS-9901 — GS-9901 tablets administered orally

SUMMARY:
This study will evaluate the safety and tolerability of GS-9901 monotherapy in adults with follicular lymphoma (FL), marginal zone lymphoma (MZL), chronic lymphocytic leukemia (CLL), or small lymphocytic lymphoma (SLL). The study will also characterize the pharmacokinetic (PK) profile of GS-9901, determine the appropriate dosing regimen of GS-9901 for use in future clinical trials, and to evaluate the efficacy of GS-9901 monotherapy in adults with FL, MZL, CLL, or SLL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FL, MZL, SLL, or CLL (meeting International Workshop on CLL [IWCLL] Criteria, 2008) as documented by medical records and with histology based on criteria established by the World Health Organization

  * FL Grades 1, 2, or 3a
  * SLL with absolute lymphocyte count of < 5 x 10^9/L at initial diagnosis
  * MZL (splenic, nodal, or extra-nodal)
* Prior treatment for FL or CLL/SLL with ≥ 1 prior chemotherapy-based or immunotherapy-based regimen with no approved therapies available
* Presence of radiographically measurable lymphadenopathy or extra nodal lymphoid malignancy
* All acute toxic effects of any prior antitumor therapy resolved to Grade ≤1 before the start of study therapy (with the exception of alopecia [Grade 1 or 2 permitted], or bone marrow parameters [any of Grade 1, 2, or 3 permitted)
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Able to provide written informed consent

Exclusion Criteria:

* History of lymphoid malignancy other than FL, MZL, SLL, or CLL
* History of myelodysplastic syndrome
* History of a non-lymphoid malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for ≥ 1 year prior to start of study therapy, or any other cancer that has been in complete remission for ≥ 5 years
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of start of study therapy
* Ongoing drug-induced pneumonitis
* Ongoing inflammatory bowel disease
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* History of prior therapy with any inhibitor of serine/threonine kinase (AKT), Bruton tyrosine kinase (BTK), Janus kinase (JAK), mammalian target of rapamycin (mTOR), phosphatidylinositol 3-kinase (PI3K), or spleen tyrosine kinase (SYK)
* Ongoing immunosuppressive therapy, including systemic corticosteroids for treatment of lymphoid malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) and clinical laboratory abnormalities defined as dose limiting toxicities (DLTs) | Up to 28 days
  Overall safety profile will be characterized by number of participants experiencing adverse events or laboratory abnormalities.

SECONDARY OUTCOMES:
Occurrence of AEs and clinical laboratory abnormalities not defined as DLTs | Up to 2 years
  Overall safety profile will be characterized by number of participants experiencing adverse events or laboratory abnormalities.
Overall response rate | Up to 2 years
  Overall response rate (ORR) is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR).
Progression-free survival | Up to 2 years
  Progression-free survival (PFS) is defined as the interval from the start of study therapy to the earlier of the first documentation of definitive disease progression or death from any cause.
Duration of response | Up to 2 years
  Duration of response (DOR) is defined as the interval from the first documentation of CR or PR to the earlier of the first documentation of definitive disease progression or death from any cause.
PK profile of GS-9901 | Predose and 0.5, 1, 1.5, 2, 3, 4, 6, and 24 hours postdose on Days 1 and 15; predose and 1.5 hours postdose on Days 29, 43, 85, and 169
  This endpoint will measure the plasma PK profile of GS-9901. The following parameters will be measured:
  * Cmax: maximum observed concentration of drug in plasma
  * AUCtau: concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Adewoye, MD, Study Director — Gilead Sciences
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - Cancer Care Center of Fresno, Fresno, California
  - Innovative Clinical Research Institute, Whittier, California
  - Cancer Center Central Connecticut, Southington, Connecticut
  - Lombardi Cancer Center-Georgetown University, Washington D.C., District of Columbia
  - Northwest Medical Specialties, Tacoma, Washington